CLINICAL TRIAL: NCT00826878
Title: A Phase 1b/2a Open-Label Study to Evaluate the Safety and Activity of Once Daily Oral Administration of Tivozanib (AV-951) in Subjects With Non-Small Cell Lung Cancer
Brief Title: An Open-Label Study of QD Oral Administration of Tivozanib (AV-951) in Subjects With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-08-105
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: tivozanib; AV-951
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tivozanib (AV-951) (Experimental)
  Interventions: Drug: Tivozanib (AV-951)

INTERVENTIONS:
Drug: Tivozanib (AV-951) — Subjects will receive 1.0 or 1.5 mg tivozanib (AV-951) once daily continuously beginning on Day 1 for 4 weeks. One cycle will be defined as 4 weeks of treatment. Cycles will be repeated every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Minimum of 8 weeks (2 consecutive dosing cycles), if tolerated.

SUMMARY:
This is a standard Phase 1b and 2a, multi-center, study design that will examine the safety, tolerability, and maximum tolerated dose of tivozanib (AV-951) with this dosing schedule, as well as overall response rate of tivozanib (AV-951) administration in NSCLC.

DETAILED DESCRIPTION:
The Phase 2a portion of the study was not conducted

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, of either sex and of any race.
2. Histologically or cytologically confirmed NSCL.
3. Stage IIIB (with malignant pleural effusion) or stage IV or recurrent disease.
4. Subjects that have recurred or progressed following standard therapy or failed standard therapy; or subjects that are not candidates for or unwilling to undergo standard therapy.
5. Disease that is currently not amenable to curative surgical intervention, due to either non-resectability of the tumor or medical contraindications.
6. Prior VEGF directed therapy
7. Prior chemotherapy
8. At least 4 weeks since prior immunotherapy (eg, IL-2, IFN, etc.) or biological therapy (eg, MABs) prior to the first dose of study drug.
9. At least 1 week since prior treatment with warfarin, acenocoumarol, fenprocoumon, or similar agents.
10. At least 4 weeks since prior systemic hormonal therapy.
11. At least 2 weeks since prior use of herbal preparations/supplements.
12. At least 2 weeks since prior treatment with CYP3A4 inducers or inhibitors.
13. At least 2 weeks since prior radiotherapy to ≤25% of bone marrow, or at least 4 weeks since prior radiotherapy to > 25% of bone marrow.
14. Measurable or evaluable disease; subjects enrolled in the Phase 2a study must have measurable disease by RECIST criteria.
15. ECOG performance 0-1 and life expectancy ≥ 3 months.
16. Ability to give written informed consent.

Exclusion Criteria:

1. Subjects with central lung lesions involving major blood vessels.
2. Primary CNS malignancies or symptomatic CNS metastases; subjects with previously treated brain metastasis will be allowed if the brain metastasis have been stable without steroid treatment for at least 3 months following prior treatment (radiotherapy or surgery).
3. Hematologic malignancies (including leukemia in any form, lymphoma, and multiple myeloma).
4. Hematologic abnormalities:
5. Serum chemistry abnormalities:
6. Significant cardiovascular disease
7. Subjects with delayed healing of wounds, active gastric ulcers, or unhealed bone fractures.
8. Serious/active infection or infection requiring parenteral antibiotics.
9. Inadequate recovery from any prior surgical procedure or major surgical procedure within 6 weeks prior to administration of first dose of study drug.
10. Inability to comply with protocol requirements.
11. History of ≥ Grade 2 hemoptysis within 6 months prior to administration of first dose of study drug; ongoing bleeding (hemoptysis, hematemesis, hematochezia or melena) or history of clinically significant bleeding within 6 months prior to administration of first dose of study drug.
12. Cerebrovascular accident within 12 months prior to administration of first dose of study drug, or peripheral vascular disease with claudication on walking less than 1 block.
13. Deep venous thrombosis or pulmonary embolus within 6 months prior to administration of first dose of study drug.
14. Subjects with a "currently active" second primary malignancy other than non-melanoma skin cancers or nonmetastatic prostate cancer. Subjects are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy and have been disease free for >2 years.
15. If female, pregnant or lactating.
16. No childbearing potential or the use of effective contraception by all fertile male and female subjects during the study and for 30 days after the last dose of study drug. All subjects must agree to use a highly effective method of contraception (including their partner).
17. Known concomitant genetic or acquired immune suppression disease such as HIV.
18. Inadequate recovery from prior antineoplastic therapy.
19. Life-threatening illness or organ system dysfunction compromising safety evaluation.
20. Psychiatric disorder, altered mental status precluding informed consent or necessary testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Ph1b: To determine the safety, tolerability, and MTD of tivozanib (AV-951) administered orally QD in subjects with NSCLC | 4 weeks (1 cycle)
Ph2a: To determine the ORR of tivozanib (AV-951) administered orally once daily in subjects with NSCLC with no prior anti-angiogenic therapy | 8 weeks (2 cycles)

SECONDARY OUTCOMES:
Ph1b: To evaluate the PK of tivozanib (AV-951) administered orally QD | 8 weeks (2 cycles)
Ph1b: To evaluate the preliminary antineoplastic activity of tivozanib (AV-951) administered orally QD | 8 weeks (2 cycles)
Ph2a: To determine the duration of complete and partial responses and time to disease progression (TTP) for subjects treated with tivozanib (AV-951) | 8 weeks (2 cycles)
Ph2a: To determine the safety and tolerability of tivozanib (AV-951) administered orally once a day | 4 weeks (1 cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Jac, M.D., Study Director — AVEO Pharmaceuticals, Inc.; Jimmy Hwang, MD, Principal Investigator — Georgetown University; Chao Huang, MD, Principal Investigator — University of Kansas; Naiyer Rizvi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Georgetown University, Washington D.C., District of Columbia
  - Kansas University Medical Center, Kansas City, Kansas
  - Memorial Sloan-Kettering, New York, New York